CLINICAL TRIAL: NCT01257061
Title: Unicentric Comparing Effectiveness Superiority of to Clemastine Fumarate 1, 0 mg/g + Dexamethasone 0, 5 mg/g to Dexchlorpheniramine Maleate 10 mg/g in Eczema Treatment.
Brief Title: Effectiveness of Clemastine Fumarate + Dexamethasone Compared to Dexchlorpheniramine Maleate in Eczema Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DECEMS1010
Record Dates: First submitted 2010-11-29; First posted 2010-12-09 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Eczema
Keywords: Dermatitis; Dermatitis, Atopic
MeSH Terms: conditions — Eczema; Dermatitis; Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Clemastine fumarate 1,0 mg/g + dexamethasone 0,5/g
  Interventions: Drug: Group 1
- Group 2 (Active Comparator): Dexchlorpheniramine maleate 10 mg/g
  Interventions: Drug: Group 2

INTERVENTIONS:
Drug: Group 1 — Clemastine fumarate 1,0 mg/g + dexamethasone 0,5/g applied 2 times / day at lesion
  Arms: Group 1
Drug: Group 2 — Dexchlorpheniramine maleate 10 mg/g applied 2 times / day at lesion
  Arms: Group 2

SUMMARY:
Atopic dermatitis is a recurrent pruritic skin disorder which has a significant morbidity and impaired quality of life due specially pruritus and physical visible skin lesions. The propose of this trial is evaluate the effectiveness of clemastine fumarate 1, 0 mg/g + dexamethasone 0, 5 mg/g compared to dexchlorpheniramine maleate 10 mg/g in eczema treatment.

DETAILED DESCRIPTION:
Study design:

• Double blinded, superiority, prospective parallel-group, intend to treat trial.

Study design:

* Experiment duration: 22 days
* 2 visits (days 1,7,15 and 22)
* Reducing Eczema Area and severity index evaluation
* Adverse events evaluation

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be able to understand the study procedures agree to participate and give written consent.
2. Patients with acute or sub-acute eczema.
3. Presence of symmetric lesions to compare on side to the other.

Exclusion Criteria:

1. Pregnancy or risk of pregnancy.
2. Lactation
3. Use of anti-inflammatory or immunosuppressive drugs (last 30 days prior to the study).
4. Sunlight over exposure in the last 15 days.
5. Any pathology or past medical condition that can interfere with this protocol.

Ages: 5 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 310 (Actual)
Dates: Start 2012-09-06 (Actual); Primary Completion 2013-04-30 (Actual); Study Completion 2013-08-02 (Actual)

PRIMARY OUTCOMES:
Reduction / improvement of signs and symptoms | DAY 22
  The reduction of signs an symptoms will be evaluated by OSAAD index.

SECONDARY OUTCOMES:
Adverse Events Evaluation | DAY 22
  Adverse events will be collected and followed in order to evaluate safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Addor, MD, Principal Investigator — Medcin Instituto da Pele; Felipe Pinho, MD, Study Director — EMS
Locations (1):
- Medcin instituto da Pele, Osasco, São Paulo, Brazil